CLINICAL TRIAL: NCT06302660
Title: Profiling Microbiome Associated Metabolic Pathways in Oesophageal Cancer Survivors
Acronym: MAPLES
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); West Hertfordshire Teaching Hospitals NHS Trust (Unknown); Barking, Havering and Redbridge University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22/LO/0169
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Oesophageal Cancer; Quality of Life; Bacterial Overgrowth
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Breath Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oesophageal adenocarcinoma survivors: 100 disease free survivors who underwent multimodality treatment for oesophageal adenocarcinoma and are >1 year post oesophagectomy
  Interventions: Diagnostic Test: Breath test; Diagnostic Test: Saliva sample; Diagnostic Test: Blood sample; Diagnostic Test: Urine sample; Diagnostic Test: Stool sample; Diagnostic Test: Health-related Quality of life questionnaires

INTERVENTIONS:
Diagnostic Test: Breath test — Participants will attend an outpatient clinic, fasted for at least 4 hours for collection of breath.
Diagnostic Test: Saliva sample — Participants will attend an outpatient clinic, fasted for at least 4 hours for collection of saliva.
Diagnostic Test: Blood sample — Participants will attend an outpatient clinic, fasted for at least 4 hours for collection of blood.
Diagnostic Test: Urine sample — Participants will attend an outpatient clinic, fasted for at least 4 hours for collection of urine.
Diagnostic Test: Stool sample — Participants will attend an outpatient clinic, fasted for at least 4 hours for collection of stool.
Diagnostic Test: Health-related Quality of life questionnaires — Participants will attend an outpatient clinic and complete validated healthy-related quality-of-life questionnaires.

SUMMARY:
The goal of this observational study is to learn about long term symptoms in oesophageal cancer survivors. The main question it aims to answer is are:

* Study the changes in gut bacteria by examining saliva, stool and blood.
* Investigate the products of bacteria in breath to develop a non-invasive breath test to detect the changes in gut bacteria.
* Develop new strategies to treat this change and trial new treatments to improve quality- of-life in oesophageal cancer survivors.

Participants will attend an outpatient clinic, fasted for at least 4 hours for collection of breath, saliva, blood, urine, stool and complete validated healthy-related quality-of-life questionnaires.

Researchers will compare symptomatic and asymptomatic participants to detect the changes stated above.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-90 years
* Patients who underwent oesophagectomy for oesophageal adenocarcinoma with curative intent
* Disease free patients (CT with no evidence of recurrence within last 6 months or more than 5 years post oesophageal resection)
* Patients more than 1 year post oesophageal resection

Exclusion Criteria:

* Patients with Siewert III gastro-oesophageal junctional tumours
* Patients with evidence of disease recurrence
* Patients who are unable or unwilling to provide informed written consent
* Patients who have received antibiotic therapy within the last 4 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disease free survivors who underwent curative treatment for oesophageal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Identify microbiome dysbiosis in saliva associated with long-term functional symptoms. | 24 months
  Metagenomic sequencing of saliva samples.
Identify microbiome dysbiosis in stool associated with long-term functional symptoms. | 24 months
  Metagenomic sequencing of stool samples.

SECONDARY OUTCOMES:
Identify underlying metabolic pathways associated with microbiome derived metabolites. | 36 months
  Bioinformatic multi-omic pathway analysis.
Develop a breath test to detect volatile biomarkers associated with microbiome dysbiosis. | 36 months
  Gas Chromatography-Mass Spectrometry (GC-MS) will be used to identify the levels (measured in parts per billion, ppb) of certain microbiome-derived VOCs in breath.
Propose a strategy for treatment of long-term symptoms in oesophageal adenocarcinoma survivors. | 36 months
  Identify therapeutic targets and interventions to manipulate dysbiotic microbiota

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Barking, Havering and Redbridge University Hospitals NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - West Hertfordshire NHS Teaching Hospitals, London